CLINICAL TRIAL: NCT02982187
Title: A Randomized, Open-label, Cross-over, Placebo-device Study Investigating Critical and Over All Errors, Training/Teaching Time, and Preference Attributes of the ELLIPTA Dry Powder Inhaler (DPI) as Compared to HANDIHALER DPI Used in Combination With Either DISKUS DPI or TURBUHALER DPI, in Adult Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Clinical Study Assessing Critical Errors, Training/Teaching Time, and Preference Attributes of the ELLIPTA® Dry Powder Inhaler, in Comparison to Combinations of Dry Powder Inhalers Used to Provide Triple Therapy, in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 206215
Record Dates: First submitted 2016-12-01; First posted 2016-12-05 (Estimated); Results first posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: HANDIHALER; ELLIPTA; TURBUHALER; DISKUS; COPD; critical error; inhaler preference
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Sub-study 1 : ELLIPTA followed by DISKUS+ HANDIHALER +PQ1 (Experimental): In this sequence, subjects will be randomized to use ELLIPTA inhaler in period 1 and then DISKUS + HANDIHALER in period 2. At the end of Visit 1, subjects will complete version 1 of the PQ (PQ1)
  Interventions: Device: Placebo ELLIPTA; Device: Placebo DISKUS; Device: Placebo HANDIHALER; Other: PQ1
- Sub-study 1 : DISKUS + HANDIHALER followed by ELLIPTA+PQ2 (Experimental): In this sequence, subjects will be randomized to use DISKUS + HANDIHALER in period 1 and then ELLIPTA in period 2. At the end of Visit 1, subjects will complete version 2 of the PQ (PQ2)
  Interventions: Device: Placebo ELLIPTA; Device: Placebo DISKUS; Device: Placebo HANDIHALER; Other: PQ2
- Sub-study 1 : ELLIPTA followed by DISKUS+ HANDIHALER +PQ2 (Experimental): In this sequence, subjects will be randomized to use ELLIPTA inhaler in period 1 and then DISKUS + HANDIHALER in period 2. At the end of Visit 1, subjects will complete PQ2
  Interventions: Device: Placebo ELLIPTA; Device: Placebo DISKUS; Device: Placebo HANDIHALER; Other: PQ2
- Sub-study 1 : DISKUS + HANDIHALER followed by ELLIPTA+PQ1 (Experimental): In this sequence, subjects will be randomized to use DISKUS + HANDIHALER in period 1 and then ELLIPTA in period 2. At the end of Visit 1, subjects will complete PQ1
  Interventions: Device: Placebo ELLIPTA; Device: Placebo DISKUS; Device: Placebo HANDIHALER; Other: PQ1
- Substudy 2: ELLIPTA followed by TURBUHALER + HANDIHALER +PQ3 (Experimental): In this sequence, subjects will be randomized to use ELLIPTA inhaler in period 1 and then TURBUHALER + HANDIHALER in period 2. At the end of Visit 1, subjects will complete version 3 of the PQ (PQ3)
  Interventions: Device: Placebo ELLIPTA; Device: Placebo TURBUHALER; Device: Placebo HANDIHALER; Other: PQ3
- Substudy 2: TURBUHALER + HANDIHALER followed by ELLIPTA+PQ4 (Experimental): In this sequence, subjects will be randomized to use TURBUHALER + HANDIHALER inhaler in period 1 and then ELLIPTA in period 2. At the end of Visit 1, subjects will complete version 4 of the PQ (PQ4)
  Interventions: Device: Placebo ELLIPTA; Device: Placebo TURBUHALER; Device: Placebo HANDIHALER; Other: PQ4
- Substudy 2: ELLIPTA followed by TURBUHALER + HANDIHALER +PQ4 (Experimental): In this sequence, subjects will be randomized to use ELLIPTA inhaler in period 1 and then TURBUHALER + HANDIHALER in period 2. At the end of Visit 1, subjects will complete PQ4
  Interventions: Device: Placebo ELLIPTA; Device: Placebo TURBUHALER; Device: Placebo HANDIHALER; Other: PQ4
- Substudy 2: TURBUHALER + HANDIHALER followed by ELLIPTA+PQ3 (Experimental): In this sequence, subjects will be randomized to use TURBUHALER + HANDIHALER inhaler in period 1 and then ELLIPTA in period 2. At the end of Visit 1, subjects will complete PQ3
  Interventions: Device: Placebo ELLIPTA; Device: Placebo TURBUHALER; Device: Placebo HANDIHALER; Other: PQ3

INTERVENTIONS:
Device: Placebo ELLIPTA — It is a dry powder inhaler device that can hold two individual blisters: one placebo strip containing lactose monohydrate and a second placebo strip containing lactose monohydrate blended with magnesium stearate.
Device: Placebo DISKUS — It is a placebo dry powder inhaler with one blister strip containing lactose monohydrate.
  Arms: Sub-study 1 : DISKUS + HANDIHALER followed by ELLIPTA+PQ1; Sub-study 1 : DISKUS + HANDIHALER followed by ELLIPTA+PQ2; Sub-study 1 : ELLIPTA followed by DISKUS+ HANDIHALER +PQ1; Sub-study 1 : ELLIPTA followed by DISKUS+ HANDIHALER +PQ2
Device: Placebo TURBUHALER — It is a placebo dry powder inhaler containing lactose monohydrate.
  Arms: Substudy 2: ELLIPTA followed by TURBUHALER + HANDIHALER +PQ3; Substudy 2: ELLIPTA followed by TURBUHALER + HANDIHALER +PQ4; Substudy 2: TURBUHALER + HANDIHALER followed by ELLIPTA+PQ3; Substudy 2: TURBUHALER + HANDIHALER followed by ELLIPTA+PQ4
Device: Placebo HANDIHALER — Placebo capsules contain lactose monohydrate in the form of powder for oral inhalation, to be used with HANDIHALER device.
Other: PQ1 — Consists of 2 questions to assess subjects' preference of device attributes and dosing regimens. The 4 versions of the questionnaire ask the same questions, but differ in the ordering of inhalers in their responses.
  Arms: Sub-study 1 : DISKUS + HANDIHALER followed by ELLIPTA+PQ1; Sub-study 1 : ELLIPTA followed by DISKUS+ HANDIHALER +PQ1
Other: PQ2 — Consists of 2 questions to assess subjects' preference of device attributes and dosing regimens. The 4 versions of the questionnaire ask the same questions.
  Arms: Sub-study 1 : DISKUS + HANDIHALER followed by ELLIPTA+PQ2; Sub-study 1 : ELLIPTA followed by DISKUS+ HANDIHALER +PQ2
Other: PQ3 — Consists of 2 questions to assess subjects' preference of device attributes and dosing regimens. The 4 versions of the questionnaire ask the same questions.
  Arms: Substudy 2: ELLIPTA followed by TURBUHALER + HANDIHALER +PQ3; Substudy 2: TURBUHALER + HANDIHALER followed by ELLIPTA+PQ3
Other: PQ4 — Consists of 2 questions to assess subjects' preference of device attributes and dosing regimens. The 4 versions of the questionnaire ask the same questions.
  Arms: Substudy 2: ELLIPTA followed by TURBUHALER + HANDIHALER +PQ4; Substudy 2: TURBUHALER + HANDIHALER followed by ELLIPTA+PQ4

SUMMARY:
This is a randomized, multi-centre, open-label, placebo-device, cross-over study, with a 2x2 complete block design in subjects with chronic obstructive pulmonary disease (COPD) to assess the benefits of delivering triple therapy using a single ELLIPTA dry powder inhaler (DPI) (closed triple therapy) versus delivering triple therapy using two different types of DPI (open triple therapy). The primary objective of the study is to evaluate the proportion of COPD subjects who make critical errors when using a single ELLIPTA DPI versus those using combinations of DISKUS® with HANDIHALER®, or TURBUHALER® with HANDIHALER. At Visit 1, all subjects will demonstrate the use of ELLIPTA DPI, and HANDIHALER DPI in combination with either DISKUS DPI (in sub-study 1) or TURBUHALER DPI (in sub-study 2), based on the treatment sequences. At the end Visit 1, subjects will complete the inhaler preference questionnaire (PQ). There is no active treatment and subjects will continue to take their own prescribed COPD medication for the duration of the study. ELLIPTA and DISKUS are registered trademarks of the GSK group of companies; TURBUHALER is a registered trademark of AstraZeneca and HANDIHALER is a registered trademark of Boehringer Ingelheim Pharma GmbH & Co. KG.

ELIGIBILITY:
Inclusion Criteria

* Age >=40 years at Visit 1
* Diagnosis of COPD with a documented history of COPD, in accordance with the definition by the European Respiratory Society.
* Current COPD Therapy: Currently receiving maintenance therapy with a fixed dose combination of a long-acting beta 2-agonist (LABA) and inhaled corticosteroid (ICS). Subject may also be receiving long-acting muscarinic antagonist (LAMA; also known as a long-acting anti-cholinergic). Subjects must be able to continue using their currently prescribed COPD maintenance inhaler therapy throughout the study and as needed short acting beta-adrenergic agonist (SABA) and/or short acting muscarinic antagonist (SAMA) for rescue use.
* Has been on current maintenance ICS/LABA COPD treatment for at least 4 weeks prior to V0 and evaluated as unlikely to change treatment within 4 weeks of Visit 1.
* Current or former (defined as subjects who have quit smoking for at least 3 months prior to V0/V1) cigarette smokers with a >10 pack-year smoking history (Number of pack years=[number of cigarettes per day ÷ 20] x number of years smoked [e.g., 10 pack-years is equal to 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years]).
* Males or females who are not pregnant or not planning a pregnancy during the study or not lactating
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria

* Subjects with a current diagnosis of asthma. Subjects with a prior history of asthma are eligible if they have a current diagnosis of COPD.
* Subjects who used any ELLIPTA inhaler (participated in a clinical study of GW685698, GW642444, GSK573719 [fluticasone furoate, vilanterol, umeclidinium bromide], or any combination thereof, or placebo in an ELLIPTA inhaler study) within 24 months prior to Visit 0.
* Subjects who used any capsule system inhaler (e.g. Spiriva HANDIHALER, SEEBRI®/ULTIBRO® BREEZHALER®, or participated in a clinical studies of these, including placebo inhalers) within 24 months prior to Visit 0. SEEBRI, ULTIBRO, and BREEZHALER are registered trademarks of Novartis AG.
* Dependent on which sub-study a subject is included on they should not have any recent experience, within 24 months of V 0 of the following inhaler for the sub study included on: Sub Study 1: DISKUS inhaler (e.g., Seretide DISKUS or placebo DISKUS) and Sub Study 2:TURBUHALER (e.g. Symbicort TURBUHALER or placebo TURBUHALER)
* Subjects with a known or suspected alcohol or drug abuse at Visit 1 which in the opinion of the investigator could interfere with the subject's proper completion of the protocol requirement
* A history of hypersensitivity to any components of the study inhaler (e.g., lactose, magnesium stearate). In addition, subjects with a history of severe milk protein allergy that, in the opinion of the study physician, contraindicates participation will also be excluded.
* Subjects who have received an investigational drug and/or medical device within 30 days of entry into this study (Screening/Visit 1), or within five drug half-lives of the investigational drug, whichever is longer
* In the opinion of the investigator, any subject who is unable to read and/or would not be able to complete a questionnaire and understand verbal instructions.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2016-12-30 (Actual); Primary Completion 2017-06-19 (Actual); Study Completion 2017-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Netherlands (3):
  - GSK Investigational Site, Enschede
  - GSK Investigational Site, Nijverdal
  - GSK Investigational Site, Rotterdam
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van der Palen J, Moeskops-van Beurden W, Dawson CM, James WY, Preece A, Midwinter D, Barnes N, Sharma R. A randomized, open-label, single-visit, crossover study simulating triple-drug delivery with Ellipta compared with dual inhaler combinations in patients with COPD. Int J Chron Obstruct Pulmon Dis. 2018 Aug 21;13:2515-2523. doi: 10.2147/COPD.S169060. eCollection 2018. PMID 30174421

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a randomized, multi-center, open-label, cross-over study comparing Placebo ELLIPTA Dry Power Inhaler (DPI) with either Placebo DISKUS DPI + Placebo Handihaler or Placebo Turbuhaler plus Placebo Handihaler to assess correct inhaler use. A total of 5 centers, 3 in the Netherlands and 2 in the United Kingdom participated in the study.
Pre-assignment Details: A total of 160 participants were screened. Eighty were assigned to sub-study 1 and 80 to sub-study 2 according to naivety to inhalers in each sub-study. One participant in sub-study 2 withdrew consent prior to device assessment. Therefore 80 par in sub-study 1 and 79 par in sub-study 2 are included in the intent to treat population.
Groups:
- ELLIPTA/DISKUS+HandiHaler/Q1: Participants received placebo via ELLIPTA in period 1 and DISKUS + HandiHaler in period 2, followed by preference questionnaire (PQ) 1. There was no active treatment and participants continued to take their own prescribed COPD medication for the duration of the study.
- ELLIPTA/DISKUS+HandiHaler/Q2: Participants received placebo via ELLIPTA in period 1 and DISKUS + HandiHaler in period 2, followed by PQ2. There was no active treatment and participants continued to take their own prescribed COPD medication for the duration of the study.
- DISKUS+HandiHaler/ELLIPTA/Q1: Participants received placebo via DISKUS + HandiHaler in period 1 and ELLIPTA in period 2, followed by PQ1 respectively. There was no active treatment and participants continued to take their own prescribed COPD medication for the duration of the study.
- DISKUS+HandiHaler/ELLIPTA/Q2: Participants received placebo via DISKUS + HandiHaler in period 1 and ELLIPTA in period 2, followed by PQ2. There was no active treatment and participants continued to take their own prescribed COPD medication for the duration of the study.
- ELLIPTA/Turbuhaler+HandiHaler/Q3: Participants received placebo via ELLIPTA in period 1 and Turbuhaler + HandiHaler in period 2, followed by PQ3. There was no active treatment and participants continued to take their own prescribed COPD medication for the duration of the study.
- ELLIPTA/Turbuhaler+HandiHaler/Q4: Participants received placebo via ELLIPTA in period 1 and Turbuhaler + HandiHaler in period 2, followed by PQ4. There was no active treatment and participants continued to take their own prescribed COPD medication for the duration of the study.
- Turbuhaler+HandiHaler/ELLIPTA/Q3: Participants received placebo via Turbuhaler + HandiHaler in period 1 and ELLIPTA in period 2, followed by PQ3. There was no active treatment and participants continued to take their own prescribed COPD medication for the duration of the study.
- Turbuhaler+HandiHaler/ELLIPTA/Q4: Participants received placebo via Turbuhaler + HandiHaler in period 1 and ELLIPTA in period 2, followed by PQ4. There was no active treatment and participants continued to take their own prescribed COPD medication for the duration of the study.
Period: Overall Study
Arm/Group | ELLIPTA/DISKUS+HandiHaler/Q1 | ELLIPTA/DISKUS+HandiHaler/Q2 | DISKUS+HandiHaler/ELLIPTA/Q1 | DISKUS+HandiHaler/ELLIPTA/Q2 | ELLIPTA/Turbuhaler+HandiHaler/Q3 | ELLIPTA/Turbuhaler+HandiHaler/Q4 | Turbuhaler+HandiHaler/ELLIPTA/Q3 | Turbuhaler+HandiHaler/ELLIPTA/Q4
Started | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20
Completed | 20 | 20 | 20 | 20 | 20 | 20 | 19 | 20
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Population comprised of all randomized participants who made at least one critical error assessment from one treatment option device. One participant withdrew consent prior to device assessment in Sub-study 2 and only 79 participants were included in Intent-to-Treat Population.
Groups:
- Sub Study 1: ELLIPTA vs DISKUS + HandiHaler: Participants received placebo via one of the following devices: ELLIPTA® DPI or DISKUS® DPI in combination with HANDIHALER® DPI based on the following four sequences. The sequences also include the preference questionnaire version: A (ELLIPTA in period 1 and DISKUS + HandiHaler in period 2,followed by PQ1), B (DISKUS + HandiHaler in period 1 and ELLIPTA in period 2,followed by PQ2), C (ELLIPTA in period 1 and DISKUS + HandiHaler in period 2, followed by PQ2), D (DISKUS + HandiHaler in period 1 and ELLIPTA in period 2, followed by PQ1) respectively. There was no active treatment and participants continued to take their own prescribed COPD medication for the duration of the study.
- Sub Study 2: ELLIPTA vs Turbuhaler + HandiHaler: Participants received placebo via one of the following devices: ELLIPTA DPI or TURBUHALER® DPI in combination with HANDIHALER DPI based on the following four sequences. The sequences also include the preference questionnaire version: : E (ELLIPTA in period 1 and Turbuhaler + HandiHaler in period 2, followed by PQ3), F (Turbuhaler + HandiHaler in period 1 and ELLIPTA in period 2, followed by PQ4), G (ELLIPTA in period 1 and Turbuhaler + HandiHaler in period 2, followed by PQ4), H (Turbuhaler + HandiHaler in period 1 and ELLIPTA in period 2, followed by PQ3) respectively. There was no active treatment and participants continued to take their own prescribed COPD medication for the duration of the study.
- Total: Total of all reporting groups
Arm/Group | Sub Study 1: ELLIPTA vs DISKUS + HandiHaler | Sub Study 2: ELLIPTA vs Turbuhaler + HandiHaler | Total
Number analyzed (Participants) | 80 | 79 | 159
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.3 (8.69) | 65.7 (8.49) | 65.0 (8.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 37 | 76
  Male | 41 | 42 | 83
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 1 | 0 | 1
  Asian - Central/South Asian Heritage | 20 | 20 | 40
  Asian - South East Asian Heritage | 1 | 0 | 1
  White - Arabic/North African Heritage | 5 | 4 | 9
  White - White/Caucasian/European Heritage | 53 | 55 | 108

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Making at Least One Critical Error After Reading the Patient Information Leaflets (PIL)
Description: Participants were provided with the relevant section of the PIL, explaining correct use, for each DPI they were to be tested on. A critical error was defined as an error that was most likely to result in no, or a significantly reduced amount, of medication being inhaled by the participant. After reading the PIL for each DPI to be tested, participants demonstrated the DPI and critical errors made by the participants while using each DPI were recorded by the Healthcare Professional (HCP) on the checklists provided. Percentage of participants making at least one critical error after reading PIL were reported.
Time Frame: Day 1
Population: Intent-to-Treat Population
Measure: Number; unit: Percentage of participants
Groups:
- Sub-study 1 : ELLIPTA: Participants were randomized to use placebo via ELLIPTA in either period 1 or 2.
- Sub-study 1 : DISKUS + HandiHaler: Participants were randomized to use placebo via DISKUS + HANDIHALER in period 1 or 2.
- Sub-study 2 : ELLIPTA: Participants were randomized to use placebo via ELLIPTA in period 1 or 2.
- Sub-study 2 : Turbuhaler + HandiHaler: Participants were randomized to use placebo via TURBUHALER + HANDIHALER in period 1 or 2.
Arm/Group | Sub-study 1 : ELLIPTA | Sub-study 1 : DISKUS + HandiHaler | Sub-study 2 : ELLIPTA | Sub-study 2 : Turbuhaler + HandiHaler
Number analyzed (Participants) | 80 | 80 | 79 | 79
Percentage of participants | 9 | 75 | 9 | 73
Statistical Analysis 1: Comparison: Sub-study 1 : ELLIPTA vs Sub-study 1 : DISKUS + HandiHaler; Sub study 1: DISKUS + HandiHaler vs ELLIPTA; Test type: Superiority; p < 0.001, stratified exact logistic model; Odds Ratio (OR) = 29.114, 95% CI 2-sided [lower limit 11.047] (The upper bound of the 95% CI could not be calculated due to the low number of events and is therefore displayed as NA.) — Odds ratio, 95% CI and P-value obtained from a stratified exact logistic model. Participant is included in the model as fixed strata, treatment option in the exact statement and period included as a fixed effect
Statistical Analysis 2: Comparison: Sub-study 2 : ELLIPTA vs Sub-study 2 : Turbuhaler + HandiHaler; Sub study 2:Turbuhaler + HandiHaler vs ELLIPTA; Test type: Superiority; p < 0.001, stratified exact logistic model; Odds Ratio (OR) = 27.744, 95% CI 2-sided [lower limit 10.512] (The upper bound of the 95% CI could not be calculated due to the low number of events and is therefore displayed as NA.) — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Percentage of Participants Making at Least One Critical Error After the First Instruction From the HCP
Description: Participants were provided with the relevant section of the PIL, explaining correct use, for each DPI they were to be tested on. A critical error was defined as an error that was most likely to result in no, or a significantly reduced amount, of medication being inhaled by the participant. After reading PIL for each DPI to be tested, participants demonstrated the DPI and errors made by the participants while using each DPI were recorded by the HCP on the checklists provided. If a participant made errors while demonstrating DPI, HCP provided instruction on the correct use of the DPI. The participant then repeated the demonstration of DPI use, and the HCP recorded the critical errors made on the checklists. Percentage of participants making at least one critical error after the first instruction from the HCP were reported.
Time Frame: Day 1
Population: Intent-to-Treat Population
Measure: Number; unit: Percentage of participants
Arm/Group | Sub-study 1 : ELLIPTA | Sub-study 1 : DISKUS + HandiHaler | Sub-study 2 : ELLIPTA | Sub-study 2 : Turbuhaler + HandiHaler
Number analyzed (Participants) | 80 | 80 | 79 | 79
Percentage of participants | 1 | 9 | 3 | 14
Statistical Analysis 1: Comparison: Sub-study 1 : ELLIPTA vs Sub-study 1 : DISKUS + HandiHaler; Sub study 1:DISKUS + HandiHaler vs ELLIPTA; Test type: Superiority; p = 0.029, stratified exact logistic model; Odds Ratio (OR) = 4.248, 95% CI 2-sided [lower limit 1.416] (The upper bound of the 95% CI could not be calculated due to the low number of events and is therefore displayed as NA.) — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Sub-study 2 : ELLIPTA vs Sub-study 2 : Turbuhaler + HandiHaler; Sub study 2:Turbuhaler + HandiHaler vs ELLIPTA; Test type: Superiority; p = 0.026, stratified exact logistic model; Odds Ratio (OR) = 3.855, 95% CI 2-sided [lower limit 1.394] (The upper bound of the 95% CI could not be calculated due to the low number of events and is therefore displayed as NA.) — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Participants Making at Least One Critical Error After the Second Instruction From the HCP
Description: Participants were provided with the relevant section of the PIL, explaining correct use, for each DPI they were to be tested on. A critical error was defined as an error that was most likely to result in no, or a significantly reduced amount, of medication being inhaled by the participant. After reading the PIL for each DPI to be tested, participants demonstrated the DPI and errors made by the participants while using each DPI were recorded by the HCP on the checklists provided. If a participant made an error while demonstrating DPI use after first instruction from the HCP, then the HCP provided instructions again on the correct use of the inhaler. The participant then demonstrated the DPI for one last time, and the HCP recorded the critical errors made on the checklists. Participants making at least one critical error after the second instruction from the HCP were reported.
Time Frame: Day 1
Population: Intent-to-Treat Population
Measure: Number; unit: Percentage of participants
Arm/Group | Sub-study 1 : ELLIPTA | Sub-study 1 : DISKUS + HandiHaler | Sub-study 2 : ELLIPTA | Sub-study 2 : Turbuhaler + HandiHaler
Number analyzed (Participants) | 80 | 80 | 79 | 79
Percentage of participants | 0 | 6 | 0 | 5
Statistical Analysis 1: Comparison: Sub-study 1 : ELLIPTA vs Sub-study 1 : DISKUS + HandiHaler; Sub study 1:DISKUS + HandiHaler vs ELLIPTA; Test type: Superiority; p = 0.400, stratified exact logistic model; Odds Ratio (OR) = 2.000, 95% CI 2-sided [lower limit 0.459] (The upper bound of the 95% CI could not be calculated due to the low number of events and is therefore displayed as NA.) — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Sub-study 2 : ELLIPTA vs Sub-study 2 : Turbuhaler + HandiHaler; Sub study 2:Turbuhaler + HandiHaler vs ELLIPTA; Test type: Superiority; p = 0.500, stratified exact logistic model; Odds Ratio (OR) = 1.732, 95% CI 2-sided [lower limit 0.397] (The upper bound of the 95% CI could not be calculated due to the low number of events and is therefore displayed as NA.) — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percentage of Participants Making at Least One Overall Error After Reading the PIL
Description: Participants were provided with the relevant section of the PIL, explaining correct use, for each DPI they were to be tested on. Overall error was defined as an error including critical and non-critical errors made by the participants while demonstrating DPI use after reading the PIL. For each DPI to be tested, overall errors including critical and non-critical errors made by the participants while demonstrating DPI use after reading the PIL were recorded by the HCP on the checklists provided. Percentage of participants making at least one overall error after reading the PIL were reported.
Time Frame: Day 1
Population: Intent-to-Treat Population
Measure: Number; unit: Percentage of participants
Arm/Group | Sub-study 1 : ELLIPTA | Sub-study 1 : DISKUS + HandiHaler | Sub-study 2 : ELLIPTA | Sub-study 2 : Turbuhaler + HandiHaler
Number analyzed (Participants) | 80 | 80 | 79 | 79
Percentage of participants | 24 | 80 | 22 | 80
Statistical Analysis 1: Comparison: Sub-study 1 : ELLIPTA vs Sub-study 1 : DISKUS + HandiHaler; Sub study 1:DISKUS + HandiHaler vs ELLIPTA; Test type: Superiority; p < 0.001, stratified exact logistic model; Odds Ratio (OR) = 24.539, 95% CI 2-sided [lower limit 9.268] (The upper bound of the 95% CI could not be calculated due to the low number of events and is therefore displayed as NA.) — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Sub-study 2 : ELLIPTA vs Sub-study 2 : Turbuhaler + HandiHaler; Sub study 2:Turbuhaler + HandiHaler vs ELLIPTA; Test type: Superiority; p < 0.001, stratified exact logistic model; Odds Ratio (OR) = 17.974, 95% CI 2-sided [lower limit 7.239] (The upper bound of the 95% CI could not be calculated due to the low number of events and is therefore displayed as NA.) — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Percentage of Participants Making at Least One Overall Error After the First Instruction From the HCP
Description: For each DPI to be tested, overall errors including critical and non-critical errors made by the participants while demonstrating DPI use after reading the PIL following first instruction from the HCP were recorded by the HCP on the checklists provided. Percentage of participants making at least one overall error after the first instruction from the HCP were reported.
Time Frame: Day 1
Population: Intent-to-Treat Population
Measure: Number; unit: Percentage of participants
Arm/Group | Sub-study 1 : ELLIPTA | Sub-study 1 : DISKUS + HandiHaler | Sub-study 2 : ELLIPTA | Sub-study 2 : Turbuhaler + HandiHaler
Number analyzed (Participants) | 80 | 80 | 79 | 79
Percentage of participants | 5 | 15 | 5 | 20
Statistical Analysis 1: Comparison: Sub-study 1 : ELLIPTA vs Sub-study 1 : DISKUS + HandiHaler; Sub study 1:DISKUS + HandiHaler vs ELLIPTA; Test type: Superiority; p = 0.067, stratified exact logistic model; Odds Ratio (OR) = 3.237, 95% CI 2-sided [lower limit 1.124] (The upper bound of the 95% CI could not be calculated due to the low number of events and is therefore displayed as NA.) — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Sub-study 2 : ELLIPTA vs Sub-study 2 : Turbuhaler + HandiHaler; Sub study 2:Turbuhaler + HandiHaler vs ELLIPTA; Test type: Superiority; p = 0.003, stratified exact logistic model; Odds Ratio (OR) = 6.357, 95% CI 2-sided [lower limit 2.219] (The upper bound of the 95% CI could not be calculated due to the low number of events and is therefore displayed as NA.) — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Percentage of Participants Making at Least One Overall Error After the Second Instruction From the HCP
Description: For each DPI to be tested, overall errors including critical and non-critical errors made by the participants while demonstrating DPI use after reading the PIL following first, and second instruction from the HCP were recorded by the HCP on the checklists provided. Percentage of participants making at least one overall error after the second instruction from the HCP were reported. These statistics are only presented when the model has successfully converged.
Time Frame: Day 1
Population: Intent-to-Treat Population
Measure: Number; unit: Percentage of participants
Arm/Group | Sub-study 1 : ELLIPTA | Sub-study 1 : DISKUS + HandiHaler | Sub-study 2 : ELLIPTA | Sub-study 2 : Turbuhaler + HandiHaler
Number analyzed (Participants) | 80 | 80 | 79 | 79
Percentage of participants | 4 | 8 | 1 | 6
Statistical Analysis 1: Comparison: Sub-study 1 : ELLIPTA vs Sub-study 1 : DISKUS + HandiHaler; Sub study 1: DISKUS + HandiHaler vs ELLIPTA; Test type: Superiority; stratified exact logistic model; These statistics were only presented when the model successfully converged. A stratified exact logistic model was used with participant included in the model as fixed strata, treatment option in the exact statement and period included as a fixed effect
Statistical Analysis 2: Comparison: Sub-study 2 : ELLIPTA vs Sub-study 2 : Turbuhaler + HandiHaler; Sub study 2:Turbuhaler + HandiHaler vs ELLIPTA; Test type: Superiority; p = 0.500, stratified exact logistic model; Odds Ratio (OR) = 1.732, 95% CI 2-sided [lower limit 0.397] (The upper bound of the 95% CI could not be calculated due to the low number of events and is therefore displayed as NA.) — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Number of Participants With Instructions (0, 1 or 2 Times) From the HCP Which Are Needed to Demonstrate Correct Inhaler Use
Description: In each sub-study, if the participant made error while demonstrating the use of the DPI after reading the PIL, the HCP demonstrated the correct usage instructions to the participant. The participant was then asked to demonstrate the DPI again. Any errors made were recorded by the HCP, and the same process was repeated one more time. In total, the HCP instructed the participants on the use of the DPI up to two times after which there were no assessment scheduled. Number of participants with instructions (0, 1 or 2) needed to demonstrate correct DPI use by the participants were reported.
Time Frame: Day 1
Population: Intent-to-Treat Population
Measure: Number; unit: Participants
Arm/Group | Sub-study 1 : ELLIPTA | Sub-study 1 : DISKUS + HandiHaler | Sub-study 2 : ELLIPTA | Sub-study 2 : Turbuhaler + HandiHaler
Number analyzed (Participants) | 80 | 80 | 79 | 79
Participants
  Number of Instructions, 0 | 61 | 16 | 62 | 16
  Number of Instructions, 1 | 15 | 52 | 13 | 47
  Number of Instructions, 2 | 1 | 6 | 3 | 11
  Failed to demonstrate correct use | 3 | 6 | 1 | 5
Statistical Analysis 1: Comparison: Sub-study 1 : ELLIPTA vs Sub-study 1 : DISKUS + HandiHaler; Sub study 1:DISKUS + HandiHaler vs ELLIPTA; Test type: Superiority; p < 0.001, Wilcoxon signed rank test; This method of analysis does not take sequence of treatment option into account
Statistical Analysis 2: Comparison: Sub-study 2 : ELLIPTA vs Sub-study 2 : Turbuhaler + HandiHaler; Sub study 2:Turbuhaler + HandiHaler vs ELLIPTA; Test type: Superiority; p < 0.001, Wilcoxon signed rank test; This method of analysis does not take sequence of treatment option into account

8. Secondary Outcome: The Median Time to Demonstrate Correct Inhaler Use (T1+T2)
Description: For each DPI being tested, the total time taken from when participant started reading the PIL until when correct use was demonstrated (that is the time required to read PIL, and two attempts for correct use of DPI following instructions provided by the HCP ) was recorded. A participant who did not demonstrate correct use at the end of the time period was censored. The median time to demonstrate correct DPI use (minutes) is taken from the Kaplan-Meier analysis. If more than 50% of the data is censored therefore the median is not applicable.
Time Frame: Day 1
Population: Intent-to-Treat Population.
Measure: Median (Full Range); unit: Minutes
Arm/Group | Sub-study 1 : ELLIPTA | Sub-study 1 : DISKUS + HandiHaler | Sub-study 2 : ELLIPTA | Sub-study 2 : Turbuhaler + HandiHaler
Number analyzed (Participants) | 80 | 80 | 79 | 79
Minutes | 2.68 [0.8 to 12.9] | 10.57 [1.5 to 42.4] | 2.58 [0.7 to 25.2] | 11.30 [3.3 to 55.8]

9. Secondary Outcome: Time Taken to Read the PIL and Demonstrate Correct Inhaler Use (T1)
Description: For each DPI being tested, the time taken from when participant started reading the PIL until when correct use was demonstrated with no need of instructions by HCP was reported. A participant who did not demonstrate correct use at the end of the time period was censored. The median time to demonstrate correct DPI use (minutes) is taken from the Kaplan-Meier analysis. If more than 50% of the data is censored therefore the median is not applicable.
Time Frame: Day 1
Population: Intent-to-Treat Population..
Measure: Median (Full Range); unit: Minutes
Arm/Group | Sub-study 1 : ELLIPTA | Sub-study 1 : DISKUS + HandiHaler | Sub-study 2 : ELLIPTA | Sub-study 2 : Turbuhaler + HandiHaler
Number analyzed (Participants) | 80 | 80 | 79 | 79
Minutes | 2.88 [0.8 to 7.2] | NA [1.5 to 19.2] — >50% of participants were censored; therefore the median is not applicable. | 2.78 [0.7 to 8.6] | NA [3.3 to 15.1] — >50% of participants were censored; therefore the median is not applicable.

10. Secondary Outcome: Time Taken to be Given Instruction by the HCP (up to 2 Times) on Use of the Inhaler and to Demonstrate Correct Inhaler Use (T2)
Description: The time in minutes from when the HCP started to instruct participant for the correct use of DPI until correct use was demonstrated including maximum of two attempts only, was recorded. A participant who did not demonstrate correct use at the end of the time period was censored. Participants who demonstrated correct use after reading the PIL (T1) were included with a time of 0 for T2. The median time to demonstrate correct DPI use (minutes) is taken from the Kaplan-Meier analysis. If more than 50% of the data is censored then the median is not applicable. Participants who demonstrated correct use after reading the PIL are included with T2=0.
Time Frame: Day 1
Population: Intent-to-Treat Population.
Measure: Median (Full Range); unit: Minutes
Arm/Group | Sub-study 1 : ELLIPTA | Sub-study 1 : DISKUS + HandiHaler | Sub-study 2 : ELLIPTA | Sub-study 2 : Turbuhaler + HandiHaler
Number analyzed (Participants) | 80 | 80 | 79 | 79
Minutes | 0.00 [0.0 to 3.3] | 2.89 [0.0 to 16.5] | 0.00 [0.0 to 6.3] | 3.12 [0.0 to 14.3]

11. Secondary Outcome: Number of Participants With Treatment Preference Based on Responses to the Preference Questionnaire, Which Considered the Number of Steps Required to Take the COPD Medication
Description: Participants demonstrated the use of ELLIPTA, and depending on the substudy DISKUS plus HandiHaler or Turbuhaler plus Handihaler. At the end of Visit 1, participants completed specific versions of the inhaler PQ (PQ1, PQ2, PQ3 or PQ4) according to the questionnaire they were randomized to. Participants assessed the inhaler preference based on the number of steps needed to take the COPD medication. Participants checked the response from the choice of ELLIPTA, DISKUS + HandiHaler (sub-study 1), Turbuhaler + Handihaler (sub-study 2) and No Preference. Number of participants with treatment preference based on responses to the preference questionnaire were reported.
Time Frame: Day 1
Population: Intent-to-Treat Population
Measure: Number; unit: Participants
Arm/Group | Sub Study 1: ELLIPTA vs DISKUS + HandiHaler | Sub Study 2: ELLIPTA vs Turbuhaler + HandiHaler
Number analyzed (Participants) | 80 | 79
Participants
  ELLIPTA | 71 | 72
  DISKUS + HandiHaler | 6 | 4
  No Preference | 3 | 3
Statistical Analysis 1: Comparison: Sub Study 1: ELLIPTA vs DISKUS + HandiHaler; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Sub Study 2: ELLIPTA vs Turbuhaler + HandiHaler; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel

12. Secondary Outcome: Number of Participants With Treatment Preference Based on Responses to the Preference Questionnaire, Which Considered Overall Treatment Preference
Description: Participants demonstrated the use of ELLIPTA, and depending on the substudy DISKUS plus HandiHaler or Turbuhaler plus Handihaler. At the end of Visit 1, participants completed specific versions of the inhaler PQ (PQ1, PQ2, PQ3 or PQ4) according to the questionnaire they were randomized to. Participants assessed the inhaler preference based on overall treatment preference. Participants checked the response from the choice of ELLIPTA, DISKUS + HandiHaler (sub-study 1), Turbuhaler + Handihaler (sub-study 2) and No Preference. Number of participants with treatment preference based on responses to the preference questionnaire were reported.
Time Frame: Day 1
Population: Intent-to-Treat Population
Measure: Number; unit: Participants
Arm/Group | Sub Study 1: ELLIPTA vs DISKUS + HandiHaler | Sub Study 2: ELLIPTA vs Turbuhaler + HandiHaler
Number analyzed (Participants) | 80 | 79
Participants
  ELLIPTA | 65 | 66
  DISKUS + HandiHaler | 7 | 3
  No Preference | 8 | 10
Statistical Analysis 1: Comparison: Sub Study 1: ELLIPTA vs DISKUS + HandiHaler; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Sub Study 2: ELLIPTA vs Turbuhaler + HandiHaler; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: Day 1
Description: Intent-to-Treat Population was used to collect Adverse Events. Since all participants received placebo as treatment, data has been clubbed for all the arms. No Serious Adverse Events or deaths were reported during this study.
Arm/Group | Sub Study 1: ELLIPTA vs DISKUS + HandiHaler | Sub Study 2: ELLIPTA vs Turbuhaler + HandiHaler
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/79
Other Adverse Events (participants affected / at risk) | 1/80 | 0/79
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sub Study 1: ELLIPTA vs DISKUS + HandiHaler (N=80) | Sub Study 2: ELLIPTA vs Turbuhaler + HandiHaler (N=79)
Laceration (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-07-18): https://cdn.clinicaltrials.gov/large-docs/87/NCT02982187/SAP_000.pdf
  • Study Protocol (2016-09-15): https://cdn.clinicaltrials.gov/large-docs/87/NCT02982187/Prot_001.pdf